CLINICAL TRIAL: NCT00366483
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple Dose Study of the Safety, Tolerability, and Pharmacokinetics of Lecozotan SR Administered Orally to Healthy Young and Elderly Subjects
Brief Title: Study Evaluating the Safety of Lecozotan SR in Healthy Young and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3098B1-130
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2007-03-16 (Estimated); Status verified 2007-03

CONDITIONS: Alzheimer Disease
Keywords: healthy young volunteers; healthy elderly volunteers; Alzheimer's disease; 5HT1A antagonist; Health; Pharmacokinetics
MeSH Terms: conditions — Alzheimer Disease | interventions — lecozotan

INTERVENTIONS:
Drug: Lecozotan SR

SUMMARY:
To assess the safety, tolerability and pharmacokinetics of single and multiple ascending oral doses of lecozotan SR in healthy young and elderly subjects.

ELIGIBILITY:
Inclusion Criteria: -Young subjects: Men aged 18 to 45 years. -Elderly subjects: Men and women ≥ 65 years of age. -Body mass index in the range of 18 to 30 kg/m2 and body weight ≥ 50 kg. -Healthy as determined by the investigator.

Exclusion Criteria: -History of any neuropsychiatric disorder. -History of drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-05

PRIMARY OUTCOMES:
The incidence of adverse events and adverse reactions will be calculated. The safety variables (vital signs, ECG parameters, and routine laboratory tests) and PK parameters will be measured throughout study period.

SECONDARY OUTCOMES:
Pharmacokinetic analysis after single and multiple dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com
Locations (1):
- Paris, France